CLINICAL TRIAL: NCT03671655
Title: Excellence in Peripheral Arterial Disease Treatment of Superficial Femoral Artery Disease With Drug-eluting Stents (XL PAD SFA DES)
Brief Title: Excellence in Peripheral Arterial Disease Treatment of Superficial Femoral Artery Disease With Drug-eluting Stents
Acronym: XLPAD DES SFA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated as we plan to start a competing study sponsored through VA CSP.
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Subhash Banerjee, Chief of Cardiology, North Texas Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dallas VA IRB #13-098
Record Dates: First submitted 2014-10-21; First posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Peripheral Vascular Diseases; Chronic Total Occlusion of Artery of the Extremities
Keywords: Superficial femoral artery; chronic total occlusion
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Drug-Eluting Stents

STUDY DESIGN:
Intervention Model Description: This is a phase 3, multi-center, randomized controlled, parallel-group study in patients with long Superficial Femoral Artery (SFA) lesions and SFA Chronic Total Occlusion (CTO), undergoing clinically indicated stent-based percutaneous revascularization .Patients will be randomized into Drug eluting stent (DES) arm (intervention) vs. Bare Metal Stent (BMS) arm (control).
Who Masked: Participant
Masking Description: The patient and study coordinator performing patient follow-up will be blinded to the allocated treatment strategy. Angiographic and US analyses will also be done blinded to study-arm allocation. Breaking the blind will be possible for any patient who develops a complication or whose clinical care requires knowledge of the study group allocation.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug-eluting stent (Experimental): Drug-eluting stent is nitinol stent coated with Paclitaxel drug Other Names: Zilver PTX stent Zilver Paclitaxel stent
  Interventions: Device: Drug-eluting stent
- Bare metal stent (Active Comparator): Bare metal stentis Nitinol alloy self expandable stent. Other Names: Bare metal stent Nitinol stent SMART Stent Viabahn stent
  Interventions: Device: Bare metal stent

INTERVENTIONS:
Device: Drug-eluting stent — Drug eluting stent which are nitinol stent coated with Paclitaxel drug
  Other Names: Zilver PTX stent; Zilver Paclitaxel stent
  Arms: Drug-eluting stent
Device: Bare metal stent — Bare metal stent is Nitinol alloy self expandable stent. Other Names: Bare metal stent Nitinol stent SMART Stent Viabahn stent
  Other Names: Bare metal stent Nitinol stent; SMART; Viabahn
  Arms: Bare metal stent

SUMMARY:
The superficial femoral artery (SFA) is frequently involved in atherosclerosis and is the most common target of lower extremity endovascular procedures performed in patients with claudication. Endovascular treatment of SFA is challenging, given its exceptional predisposition to atherosclerosis and its exposure to extreme mechanical forces of extension, compression, torsion and flexion. The SFA is located in a fibro-muscular canal, follows a tortuous course and is considered a 'hostile' location for endovascular procedures, especially stents due to the risk of stent fracture. On the other hand, durability of balloon angioplasty in the SFA is dismal (25% patency at 1 year). Therefore, Nitinol (a metal alloy of nickel and titanium) stent implantation is the mainstay of endovascular SFA interventions when balloon angioplasty (PTA) leads to sub-optimal results during a procedure. It is used in over 70% of all cases and in nearly 100% of all femoro-popliteal (FP) CTO (chronic total occlusions) and long (≥60 mm) interventions. Endovascular treatment of SFA is challenging and restenosis is the most common cause for the lack of durability of a SFA peripheral vascular interventional procedure.5 Restenosis rates of SFA bare metal (nitinol) stents or BMS at 1 year exceeds 50% for lesions ≥60 mm in length or CTO. Stent based treatment of the SFA may not offer any additional advantage for short non-CTO (<60 mm) lesions compared to PTA. In a recent study, primarily comparing drug-eluting stents (DES) to balloon angioplasty in the SFA, 12 month patency rates were 83.1% and 32.8%, respectively for DES and balloon angioplasty arms. However, there are no head-to head studies randomized studies comparing DES and BMS in the SFA. Thus, endovascular SFA intervention in patients with symptomatic PAD is an area of urgent need for high-quality evidence as volume of these procedures continues to rise exponentially in the U.S. and around the world, largely on the basis of insufficient evidence.Thus, the purpose of this study is to conduct a randomized pilot trial comparing DES and BMS for percutaneous revascularization of SFA.

DETAILED DESCRIPTION:
Current practice of SFA revascularization almost always results in use of a Nitinol (a nickel-titanium alloy) BMS. Balloon angioplasty of complex SFA lesions, such as CTO or ≥60 mm lesions is associated with >50% restenosis at 1-year and Nitinol stents have outperformed stainless-steel stents in the SFA. Debulking strategies are employed selectively and rarely as a stand-alone therapy of SFA CTO. Stent use in long SFA lesions and CTO is fraught with the risk of fracture, mechanical deformation, neo-intimal hyperplasia and thrombosis, each of which is associated with loss of patency. Repeat procedures for in-stent restenosis are technically difficult, carry a higher morbidity compared to the initial procedure and provide less symptom relief. Therefore improving the patency of the initial procedure is in the best interest of the patient and the operator. Though long SFA lesions and CTO constitute ≥50% of all SFA lesions, it is systematically under-represented in the current SFA randomized trials. Stenting has not been shown to be superior to balloon angioplasty for short (30-60 mm) SFA lesions.SFA stenting is associated with lower patency rates and is especially less durable in diabetics, who have a higher prevalence of long lesions and CTO. In one of the largest to date outcome analyses of Nitinol stents in the SFA, 56% of lesions constituted a CTO. Seventy two percent of lesions treated with stents presented with in-stent restenosis compared to 52% of lesions stented for non-CTO lesions (p<0.001). In a multivariate analysis of stent patency, presence of a long lesion or CTO was an independent adverse predictor (hazard rate or HR=5.075, 95% confidence interval or CI 2.715-9.487). It is important to note that the benefit of stents is greater for longer and more complex lesions, including SFA CTO and long (≥60 mm) lesions.

Study subjects will be recruited from the group of patients who are referred for clinically indicated endovascular treatment of SFA for claudication at the Dallas VA Medical Center and at other participating study sites. The study the investigators propose is significant because: (a) it would affect many veterans, (b) the consequences of early SFA stent failure are grave, (c) treatment of SFA lesions is challenging, and (d) outcomes after treatment of SFA lesions are poor and may be improved with DES. In summary, failure of stent patency after initial revascularization with stenting is common and carries significant morbidity. If restenosis rates of SFA stents can be reduced with DES, it could significantly improve procedural success, durability of treatment, quality of life of patients, reduce the need for repeat revascularization procedures, and potentially reduce healthcare costs.

The proposed study is a phase 3, randomized controlled, parallel-group study in patients with long SFA lesions and SFA CTO, undergoing clinically indicated stent-based percutaneous revascularization.

End points :

The primary study end point is binary restenosis, as assessed by duplex ultrasonography performed at 12 months post-procedure or earlier if clinically indicated. Binary restenosis is defined as ≥2.5 fold increase in PSVR within the stented segment and within 10 mm of its proximal and distal edges to that recorded proximal to the stented segment or by the presence of an occluded stent with no flow. Secondary endpoints included change of resting ankle-brachial index (ABI) and symptoms (Rutherford-Becker stages), at 12 months post-procedure. Patients will be asked to complete a walking impairment questionnaire (score range: 0 to 14,080) pre-intervention, and then at 12 months for the first year post-procedure.19 All analyses will be performed in a blinded fashion at the Veterans Affairs North Texas Clinical Angiographic and Ultrasound Core Laboratory and clinical adjudication and adverse events monitoring will be performed by an independent data oversight and safety monitoring board.

Statistical analysis :

The investigators calculated a priori that 55 vascular segments would be needed in each study arm to have 80% power to detect a reduction in binary restenosis from 40% in the BMS arm to 15% in the DES arm, assuming 10% attrition and an alpha of 0.05. Continuous variables will be summarized as mean ± standard deviation and compared using the t-test or the Wilcoxon rank-sum test, as appropriate. Discrete variables will be presented as frequencies and group percentages compared using the chi-square test or Fisher's Exact Test, as appropriate. Freedom from restenosis will be assessed using Kaplan-Meier curves and log-rank test. For all comparisons a two-sided probability of <0.05 will be considered statistically significant. All analyses will be performed using SAS 9.1 (SAS Institute Inc., Cary, North Carolina).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Referred for clinically indicated lower extremity angiography and peripheral arterial intervention
3. Willing and able to give informed consent. The patients must be able to comply with study procedures and follow-up.
4. Absence of allergy to both clopidogrel and aspirin
5. Negative pregnancy test or breast-feeding
6. No coexisting conditions that limit life expectancy to less than 12 months or that could affect a patient's compliance with the protocol as per the site investigator
7. Serum creatinine <2.5 mg/dL
8. Baseline hemoglobin >9 g/dl
9. Baseline platelet count >80,000/L
10. Absence of prior stroke or transient ischemic attack within 3 months
11. ≥30 days from any prior surgical or endovascular procedure

Angiographic enrollment criteria:

1. Undergoing SFA revascularization with the intention for stent implantation
2. De novo SFA lesion ≥60 mm in length by visual estimation
3. Successfully crossed de novo SFA CTO of any length by visual estimation

Exclusion Criteria:

1. SFA lesion involving <5mm of ostial SFA and/or profunda femoris artery take-off
2. SFA lesion extending below the medial femoral epicondyle
3. <1 vessel below-the knee (BTK) run-off

   -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-01; Primary Completion 2015-08-31 (Actual); Study Completion 2015-08-31 (Actual)

PRIMARY OUTCOMES:
SFA stent patency | 12 months - The study was closed due to lower than anticipated eligible participants.
  The primary endpoint is to compare the SFA stent patency (defined as peak systolic velocity ration or PSVR≥2.5) at 12 months following percutaneous revascularization of SFA with implantation of either DES or BMS, assigned randomly to each lesion.

SECONDARY OUTCOMES:
Crossing time | 12 months - The study was closed due to lower than anticipated eligible participants
  SFA CTO crossing time with wire-catheter technique versus a dedicated CTO crossing device, as per operator discretion
Procedural duration | 12 months - The study was closed due to lower than anticipated eligible participants
  Entire procedural duration from time of getting access to dilating SFA post stenting
Composite of Major Adverse Events | 12 months - The study was closed due to lower than anticipated eligible participants
  the incidence of major adverse events (composite of all cause death, non-fatal myocardial infarction, unplanned surgical revascularization of the treated limb or amputation of the treated limb) and major bleeding (defined by GUSTO trial criteria) during the 12-month study period
Ankle Brachial Index | 12 months - The study was closed due to lower than anticipated eligible participants
  Change in ABI at 12 months compared to pre-intervention value for the target limb.
Rutherford Category | 12 months - The study was closed due to lower than anticipated eligible participants
  Change in Rutherford category symptoms at 12 months compared to pre-intervention value for the target limb.
Walking Impairment Questionnaire (WIQ) | 12 months - The study was closed due to lower than anticipated eligible participants
  Change in Walking Impairment Questionnaire at 12 months compared to pre-intervention value for the target limb.
6 minute Walking Test | 12 months - The study was closed due to lower than anticipated eligible participants
  Change in 6 minute Walking Test at 12 months compared to pre-intervention value for the target limb.

CONTACTS AND LOCATIONS:
Overall Officials: Subhash Banerjee, MD, Study Chair — North Texas Veterans Health Care System, Dallas, TX
Locations (2):
- United States (2):
  - North Texas Veterans Affairs Health Care System, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scheinert D, Scheinert S, Sax J, Piorkowski C, Braunlich S, Ulrich M, Biamino G, Schmidt A. Prevalence and clinical impact of stent fractures after femoropopliteal stenting. J Am Coll Cardiol. 2005 Jan 18;45(2):312-5. doi: 10.1016/j.jacc.2004.11.026. PMID 15653033
- [Background] Rocha-Singh KJ, Jaff MR, Crabtree TR, Bloch DA, Ansel G; VIVA Physicians, Inc. Performance goals and endpoint assessments for clinical trials of femoropopliteal bare nitinol stents in patients with symptomatic peripheral arterial disease. Catheter Cardiovasc Interv. 2007 May 1;69(6):910-9. doi: 10.1002/ccd.21104. PMID 17377972
- [Background] Krankenberg H, Schluter M, Steinkamp HJ, Burgelin K, Scheinert D, Schulte KL, Minar E, Peeters P, Bosiers M, Tepe G, Reimers B, Mahler F, Tubler T, Zeller T. Nitinol stent implantation versus percutaneous transluminal angioplasty in superficial femoral artery lesions up to 10 cm in length: the femoral artery stenting trial (FAST). Circulation. 2007 Jul 17;116(3):285-92. doi: 10.1161/CIRCULATIONAHA.107.689141. Epub 2007 Jun 25. PMID 17592075
- [Background] Dake MD, Ansel GM, Jaff MR, Ohki T, Saxon RR, Smouse HB, Zeller T, Roubin GS, Burket MW, Khatib Y, Snyder SA, Ragheb AO, White JK, Machan LS; Zilver PTX Investigators. Paclitaxel-eluting stents show superiority to balloon angioplasty and bare metal stents in femoropopliteal disease: twelve-month Zilver PTX randomized study results. Circ Cardiovasc Interv. 2011 Oct 1;4(5):495-504. doi: 10.1161/CIRCINTERVENTIONS.111.962324. Epub 2011 Sep 27. PMID 21953370
- [Background] Schillinger M, Sabeti S, Loewe C, Dick P, Amighi J, Mlekusch W, Schlager O, Cejna M, Lammer J, Minar E. Balloon angioplasty versus implantation of nitinol stents in the superficial femoral artery. N Engl J Med. 2006 May 4;354(18):1879-88. doi: 10.1056/NEJMoa051303. PMID 16672699
- [Background] Banerjee S, Das TS, Abu-Fadel MS, Dippel EJ, Shammas NW, Tran DL, Zankar A, Varghese C, Kelly KC, Weideman RA, Little BB, Reilly RF, Addo T, Brilakis ES. Pilot trial of cryoplasty or conventional balloon post-dilation of nitinol stents for revascularization of peripheral arterial segments: the COBRA trial. J Am Coll Cardiol. 2012 Oct 9;60(15):1352-9. doi: 10.1016/j.jacc.2012.05.042. Epub 2012 Sep 12. PMID 22981558